CLINICAL TRIAL: NCT06184308
Title: Pilot Clinical Trial of a Home-based Program of Rehabilitation With Health Coaching to Improve Outcomes in Post-intensive Care Syndrome Patients
Brief Title: Improving Outcomes in PICS With Home-Based Program of Rehabilitation and Health Coaching
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Rodrigo Cartin-Ceba, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-006637
Record Dates: First submitted 2023-12-14; First posted 2023-12-28 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Post-Intensive Care Syndrome
MeSH Terms: conditions — postintensive care syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Piolt (Aim 1) Group: Home-Based Program of Rehabilitation and Health Coaching (Experimental): 5-10 subjects will be assigned to complete 20 minutes of Home-based Physical Rehabilitation and Health Coaching for approximately 12 weeks to test feasibility of the home-based rehabilitation program. This will be the initial phase of the study prior to RCT phase.
  Interventions: Behavioral: Health Coaching
- Home-Based Program of Rehabilitation and Health Coaching (Experimental): Subjects will complete 20 minutes of Home-based Physical Rehabilitation and Health Coaching for approximately 12 weeks.
  Interventions: Behavioral: Home-based Physical Rehabilitation; Behavioral: Health Coaching
- Usual Care (No Intervention): Subjects will receive clinical standard of care.

INTERVENTIONS:
Behavioral: Home-based Physical Rehabilitation — Six out of seven days a week, gentle flexibility practice (upper arm and shoulder movements) that can be done seated or standing and two slow walking sessions focused on balance. In addition, complete a breathing practice focused on breathing in through the nose and exhaling through the mouth.
  Arms: Home-Based Program of Rehabilitation and Health Coaching
Behavioral: Health Coaching — Study-trained nurse whom utilizes participant data to guide interactions in weekly calls.
  Arms: Home-Based Program of Rehabilitation and Health Coaching; Piolt (Aim 1) Group: Home-Based Program of Rehabilitation and Health Coaching

SUMMARY:
The purpose of this study is to gather information on the effectiveness of a home-based rehabilitation program that also includes health coaching in patients who may suffer from post-intensive care syndrome (PICS). Many patients who are admitted to a hospital ICU suffer from new or worsening symptoms related to their medical condition and ICU care. These new or worsening symptoms may persist for some time and are collectively called post-intensive care syndrome (PICS).

ELIGIBILITY:
Inclusion Criteria:

* Adults (age ≥ 18) with PICS defined as admitted to the ICU for more than 48 hours with any of the following conditions: respiratory failure of any cause requiring mechanical ventilation ≥ three days, any shock requiring vasopressors and/or inotropes, development of delirium during the ICU stay, , and cardiac arrest during the index hospital admission.
* A HABC-M-SR score > 12 points.

Exclusion Criteria:

* Any mechanical ventilation in the last two months before the index ICU admission
* ≥ 5 days in the ICU over the previous month before the index ICU admission
* Receiving hospice or palliative care
* Severe uncontrolled psychological or psychiatric disorders, e.g., schizophrenia, bipolar disorder, struggling to cope as a result of their personality disorder, uncontrolled substance abuse (alcoholism, illegal drugs) homelessness would make them unsuitable for the intervention
* A co-morbidity so severe it would prevent the patient from engaging fully in the intervention/ control, e.g., progressive cancer, anoxic brain injury, severe rheumatoid arthritis or osteoarthritis, multiple sclerosis, chronic widespread pain syndrome, previous cerebral vascular event that the patient would not be able to participate in PR
* Patients with moderate/severe cognitive impairment per medical records screening
* Inability to obtain informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2024-05-08 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Completion of home-based rehabilitation program | 12 weeks
  Total number of subjects to complete the home-based rehabilitation program per protocol
Change in health related quality of life | Baseline, 3 months
  Measured by the European Quality of Life 5 Dimensions 5 Level (EQ-5D-5L) score. Questionnaire assess 5 dimensions of health (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) on a 5 level severity scale of no problems, slight problems, moderate problems, severe problems, and unable to perform or extreme problems.

SECONDARY OUTCOMES:
Change in Anxiety and Depression | Baseline, 3 months
  Measured using the Hospital Anxiety and Depression Scale (HADS) assessing subjects feelings in the past week. Total score 0-21 with 0-7 = normal, 8-10 borderline abnormal; and 11-21 abnormal.
Change in Post-Traumatic Stress Disorder (PTSD) Symptoms | Baseline, 3 months
  Measured using the Impact of Events Scale-Revised (IES-R) to assess subjective distressing difficulties experienced in the past seven days after a specific stressful event. 22 questions with total scoring range of 0 to 88 with 24 or more indicating PTSD is a clinical concern; 33 and above represents probable diagnosis of PTSD; and 37 or more high enough to suppress immune system's functioning.
Change in cognition | Baseline, 3 months
  Measured by the Healthy Aging Brain Care (HABC)-Monitor self-reported version questionnaire to assess brain health using a scale of not all (0-1 day); several days (2-6 days); more than half the days (7-11 days); and almost daily (12-14 days). Total score range of 0 to 81 with higher scores indicating poor cognitive, functional and behavioral brain health.
Change in Daily Steps | Baseline, 3 months
  Number of daily steps taken measured by wearable devices
Change in Sedentary Time | Baseline, 3 months
  Total sedentary time in hours measured by wearable devices
Change in Physical activity | Baseline, 3 months
  Total time recorded in in light, moderate, and strenuous physical activity in hours measured by wearable devices
Change in Sleep time | Baseline, 3 months
  Total sleep time in hours measured by wearable devices
Healthcare Utilization | 3 months
  Number of hospitalizations, outpatient, and ER visits

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Cartin-Ceba, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Mayo Clinic Minnesota, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials